CLINICAL TRIAL: NCT02717702
Title: Abbott Stress-Delta Biomarkers for ACS Risk Stratification
Brief Title: Stress-Delta Biomarkers for Acute Coronary Syndrome Risk Stratification
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00056764
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ACS Patients: Subjects will be patients presenting to the Emergency Department for evaluation of ACS.

SUMMARY:
Acute Coronary Syndrome (ACS) is a serious heart condition that is a leading cause of death in America. Cardiac stress testing is currently the best test to non-invasively identify which patients might be having ACS and may need more invasive testing such as a cardiac catheterization (placing a tube in the heart) for coronary angiogram (invasive mapping of the blood vessels of the heart). However, stress tests require imaging by highly trained specialists and even then may not correctly categorize a small minority of patients being evaluated for ACS.

Advances in blood tests may now allow detection of the very early stages of heart blood vessel blockage via a simple blood test. The investigators seek to determine whether these blood tests can help to better identify patients with ACS. The study will also store any extra blood sample that may be left over for future use.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting to the ED with clinical suspicion of ACS as determined by the treating emergency physician. These include symptoms including but not limited to chest pain, pressure, or burning sensation across the precordium.
* Age 40 years or older.
* As part of their usual clinical care, the subject is scheduled to have a cardiac stress test. This includes nuclear (adenosine, regadenosine, or other adjunct with SPECT), either pharmacologic (dobutamine) or exercise (treadmill) echocardiography, or cardiac magnetic resonance imaging. Prior cardiac testing or observation unit evaluation is not an exclusion criterion.

Exclusion Criteria:

* Patient with cardiac marker diagnosis of acute myocardial infarction or who otherwise is not a candidate for a cardiac stress test.
* Evidence of serious arrhythmias or acute MI or ischemia on ECG
* Unstable vital signs: persistent (> 2 readings or over 2 hours) hypotension (systolic blood pressure < 80 mm Hg), pulse > 110 beats per minute.
* Any medical condition that would be worsened by cardiac stress
* Aortic aneurysm or dissection
* Active myocarditis or pericarditis
* Ventricular dysrhythmia or significant atrial dysrhythmia
* Severe or greater degree of aortic stenosis
* Acute or decompensated heart failure or pulmonary edema
* Pulmonary embolism
* Aortic aneurysm
* Patient is non-English speaking.
* Patient is incarcerated or a prisoner.
* Patient does not have capacity to consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants are patients presenting to the Emergency Department for evaluation of ACS.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
% Post Stress-Delta | 1 hour
  1-hour Post-Stress Troponin I - Resting Baseline Troponin I)/ Resting Baseline Troponin I
% 2-hour Stress-Delta | 2 hour
  (3-hour Post-Stress Troponin I - Resting Baseline Troponin I)/ Resting Baseline Troponin I

SECONDARY OUTCOMES:
Delta BNP values | 1hr
Delta BNP values | 2hr

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Limkakeng, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States